CLINICAL TRIAL: NCT02459002
Title: Prospective Study to Determine Impact of Early Palliative Care Consult on Quality of Life (QOL), Cancer Related Symptoms In Advanced Lung Cancer Patients
Brief Title: Prospective Study to Determine Impact of Early Palliative Care Consult on Quality of Life (QOL), Cancer Related Symptoms In Advanced Lung Cancer Patients: Thoracic Pilot Project
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0405; NCI-2019-02352 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: Advanced lung cancer; NSCLC; palliative care
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens drawn (24 mL (8 mL x 3) at the following timepoints: baseline, every 4 weeks (+ 5 days) until end of follow-up.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NSCLC - Current Palliative Care Referral Practices: Early palliative consultation impact assessment via questionnaires during a regularly scheduled clinic visit or during inpatient stay.
  Interventions: Behavioral: QOL Questionnaire
- Primary Caregiver: Caregiver satisfaction with quality of care and early palliative consultation impact assessed via questionnaires during a regularly scheduled clinic visit or during inpatient stay.
  Interventions: Behavioral: Caregiver Satisfaction Questionnaire
- NSCLC - After Early Palliative Care Consult System: Palliative consultation impact assessment via questionnaires during a regularly scheduled clinic visit or during inpatient stay.
  Interventions: Behavioral: QOL Questionnaire

INTERVENTIONS:
Behavioral: QOL Questionnaire — Participant outcomes assessed with survey
  Other Names: survey
  Groups: NSCLC - After Early Palliative Care Consult System; NSCLC - Current Palliative Care Referral Practices
Behavioral: Caregiver Satisfaction Questionnaire — Caregiver satisfaction with quality of care assessed with surveys
  Other Names: survey
  Groups: Primary Caregiver

SUMMARY:
The goal of this study is to learn about the quality of life (QOL) in participants with advanced lung cancer.

DETAILED DESCRIPTION:
Advanced lung cancer (ALC) will be assessed for participant outcomes in a sample which is prior initiation of palliative consultation and in a sample after the initiation of early palliative consultation.

Study goals are:

I. To determine the differences in participant outcomes including quality of life (QOL); symptom distress [Edmonton symptom assessment scale (ESAS)] and caregiver outcomes [Zarit Burden Interview {ZBI}, Hospital Anxiety and Depression scale(HADS) and FAMCARE] at week 12 in advanced lung cancer (ALC) patients receiving early palliative care consultation versus those who don't.

II. Identify the cellular, molecular, and immune basis for the development of symptoms in patients with ALC.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnoses of advanced NSCLC (defined as locally advanced or metastatic)
2. Have no clinical evidence of cognitive failure, as evidenced by a Memorial Delirium Assessment Score of less than or equal to 7 of 30 ⁭at the time of consent.
3. Be at least 18 years of age.
4. Be able to understand the description of the project and give written informed consent.
5. Plan to receive their cancer treatment at MD Anderson Cancer Center.
6. Individuals with advanced cancer who are able to identify a primary caregiver who also agrees to participate (in person or by telephone) in the study. A caregiver will be defined as a spouse, first degree relative, or other person designated by the patient as providing direct assistance to the patient in his/her activities of daily living.

Exclusion Criteria:

1. Patients to be excluded from the study will be those unable to complete the baseline assessment forms or to understand the recommendations for participation in this project.
2. Patients seen at the Thoracic center at UT MD Anderson Cancer Center after 8 weeks of the initial diagnosis (first cohort only - patients using the current Palliative Care referral practices prior to the implementation of the early palliative care program).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center Non-small cell lung cancer (NSCLC) patients
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2012-07-18 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Participants' QOL Assessments | Baseline till participant death or end of follow-up period, assessed every 4 weeks for approximately 12 weeks
  Impact of early palliative consultation (defined as palliative consultation within 8 weeks of initial advanced cancer diagnosis) on participant outcomes including improvement QOL [FACT-L trial outcome index [TOI] score)]. QOL assessed with FACT-L instrument, widely used to assess QOL of advanced NSCLC. FACT-L consists of 4 general & 1 lung cancer symptom-specific subscale. General subscales include physical well-being (PWB; seven items), social/family well-being (seven items), emotional well-being (five items), and functional well-being (FWB; seven items). The seven-item lung cancer subscale (LCS) assesses symptoms commonly reported by lung cancer patients (e.g., shortness of breath, loss of weight, tightness in chest). The 21-item TOI (Trial Outcome Index) is derived by adding PWB, FWB, and LCS scores. All FACT-L items are rated on five-point scales ranging from 0 for "not at all" to 4 for "very much." Higher scores are representative of better QOL or fewer symptoms.

SECONDARY OUTCOMES:
Caregiver Outcomes: FAMCARE Scale | Baseline till participant death or end of follow-up period, assessed every 4 weeks for approximately 12 weeks
  Caregiver satisfaction with quality of care assessed with FAMCARE validated 12-item survey, which measures the degree of satisfaction with health care in terms of information provided, availability of care, physical individual with advanced cancer care, and psychological care.

CONTACTS AND LOCATIONS:
Overall Officials: Siriam Yennu, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org